CLINICAL TRIAL: NCT03273088
Title: A Randomised, Two-period, Two-sequence, Single-dose and Cross-over Study in Healthy Subjects to Demonstrate Pharmacokinetic Equivalence of Altebrel (Produced by Aryogen Pharmed) and Enbrel® (the Reference Drug, Produced by Amgen Company)
Brief Title: Pharmacokinetic, Safety and Tolerability Study of Altebrel in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ARY.ETA.AJ.PH1.2016
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2017-09

CONDITIONS: Phase 1; Bioequivalence
Keywords: healthy subjects; Pharmacokinetics; etanercept; single dose; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AryoGen Pharmed etanercept (Experimental): Altebrel (etanercept prefilled syringe produced by AryoGen Pharmed Company) 25mg/0.5ml in prefilled syringe.
  Interventions: Drug: Etanercept
- Pfizer etanercept (Active Comparator): Enbrel® (etanercept prefilled syringe produced by Pfizer Company) 25mg/0.5ml in prefilled syringe.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — A single dose of etanercept (25mg/0.5ml prefilled syringe) was administered subcutaneously to healthy subjects.
  Other Names: Altebrel; Enbrel

SUMMARY:
This study aims to demonstrate pharmacokinetic (PK) similarity of biosimilar candidate Altebrel relative to etanercept reference product (Enbrel®) and evaluate safety and tolerability of Altebrel, in a crossover fashion in healthy male volunteers after administration of a single dose (25 mg) of etanercept.

The primary objective of this study is to demonstrate that the PK of Altebrel is similar to its originator, Enbrel®, as assessed by the area under the serum concentration time curve (AUC) from time 0 extrapolated to infinity (AUCinf) and the Cmax.

The secondary objectives of the study are:

To further compare the PK of Altebrel and Enbrel®. To assess the safety of Altebrel.

DETAILED DESCRIPTION:
This is a single-dose trial with one administration of each product (Altebrel and Enbrel®). Each subject participates in two treatment period, and are randomised to receive Altebrel or Enbrel® in a crossover fashion. The subjects are closely monitored during the following 24 hours (h), and are allowed to leave the site in the next morning post evaluation and blood samples are collected prior to and at the following time points after the dose: 6, 12 and 24 hours post-dose (on day 2). The subjects are requested to visit the trial site 36, 48, 60, 72, 96, 120, 144, 168, 216, 312 and 480 h after dose administration for blood sampling and evaluation of safety variable and tolerability.

Before initiation, the trial is reviewed by food and drug administration of Iran. The protocol, electronic case report form (eCRF), information for subjects and informed consent form are submitted to the ethics committees responsible for review and approval purposes, according to national regulatory guidelines.

In this study, no subject is recruited without an informed consent. All the informed consent forms which are signed by the subjects have two copies so that subjects could receive a copy of it.

This is a crossover trial with a single dose of Altebrel and Enbrel®, separated by 28 days. 34 (group A=17, group B=17) eligible subjects have been planned to enter to the study. All of whom are aged between 18 and 55 years. Subjects' randomization is done, using permuted block and subjects are assigned to treatment sequences AB or BA. Both groups receive 25 mg of either of the drugs as a single subcutaneous injection. The injection method and prefilled syringes are totally the same in both groups. The primary objective of this study is to demonstrate that the PK of Altebrel is similar to its originator, Enbrel®, as assessed by the area under the serum concentration time curve (AUC) from time 0 extrapolated to infinity (AUCinf) and the Cmax. Secondary objectives include assessment of the time to Cmax (tmax), AUC from time 0 to the last quantifiable concentration (AUClast) of Altebrel compared with Enbrel®, as well as evaluation of safety and tolerability. The safety endpoints of the trial are to evaluate the incidence of reported adverse effects, detecting changes in vital signs, clinical laboratory tests (hematologic, biochemistry, urine analysis and urine culture tests) and ECG.

Determination of sample size:

In an equivalence test of means using two one-sided tests on data from a two-period cross-over design, a total sample size of 34 achieves 81% power at a 10% significance level when the true ratio of the means is 1/0000, the coefficient of variation on the original, unlogged scale is 0/3600, and the equivalence limits of the mean ratio are 0/8000 and 1/2500.

DATA QUALITY ASSURANCE:

AryoGen pharmed Company conducts clinical trials according to procedures that incorporate the ethical principles of GCP. Accurate and reliable data collection was assured by verification and cross-check of the eCRFs against the subject's records by clinical monitors (source document verification was performed), and the maintenance of a drug-dispensing log by the center. A comprehensive validation check program was used to verify the data, and discrepancy reports were generated accordingly for resolution by the investigator.

Blinding:

This is a double-blind trial. During the clinical phase of the trial, neither the subjects nor the site personnel are aware of the identity (Altebrel and Enbrel®) of the treatments administered. However, there is an unblinded person who receives the randomisation list and dispenses the trial drugs according to the list. The unblinded person is not otherwise participate in the execution of the trial. The randomisation list determines the dispensing order of the trial products for each subject and only the randomisation number appear on the sample collection logs, as well as, on the sample aliquots delivered to the bioanalytical laboratory. Thus, the personnel responsible for analysing the PK samples are also be blinded.

Randomisation envelopes are stored in the ISF, in a locked cabinet. In a case of emergency, the code of an individual subject may be opened and the reasons for opening will be documented and the subject will be discontinued from the trial

ELIGIBILITY:
Inclusion Criteria:

* Provide written IC to participate in the trial and to comply with the trial procedures.

  2) Take written informed consent to participate in the trial and to abide by the trial restrictions.

  3) Be healthy male between the ages of 18 and 55 years. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests.

  4) Have a body mass index between 20.0 and 29.9kg/m², inclusive 5) Have Chest X ray with no evidence of current, active TB or previous (inactive) TB, general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or within 24 weeks prior to Day 1 and read by a qualified radiologist

Exclusion Criteria:

1. Being doubtful about their availability to complete the trial.
2. history and/or current presence of clinical significant atopic allergy, hypersensitivity or allergic reactions, also including known or suspected clinically relevant drug hypersensitivity to any components of the test and reference IMP formulation or comparable drugs.
3. Active or latent Tuberculosis or who have a history of Tuberculosis.
4. history of invasive systemic fungal infections or other opportunistic infections
5. systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
6. serious infection associated with hospitalisation and/or which required intravenous antibiotics
7. history of and/or current cardiac disease
8. Have received live vaccine(s) within 30 days prior to Screening or who will require live vaccine(s) between Screening and the final study visit.
9. Intake medication with a half-life > 24 h within 1 month or 5 half-lives of the medication prior to the first administration of IMP.
10. Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody. A positive test for HIV antibody.
11. History of CNS demyelinating disorders in family (MS)
12. Have a history of smoking >10 cigarettes per day

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-12-04 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUCinf) | 21 days
  AUCinf will be calculated using the equation:AUCinf= AUClast + (Clast / Kel)
Maximum serum concentration (Cmax) | 21 days
  It is obtained directly from the observed concentration-time data

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) | 21 days
  It is calculated using the linear trapezoidal rule
Time to Cmax (Tmax) | 21 days
  It is obtained directly from the observed concentration-time data

CONTACTS AND LOCATIONS:
Locations (1):
- Orchidpharmed PK/PD site, Tehrān, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee YJ, Shin D, Kim Y, Kang J, Gauliard A, Fuhr R. A randomized phase l pharmacokinetic study comparing SB4 and etanercept reference product (Enbrel(R)) in healthy subjects. Br J Clin Pharmacol. 2016 Jul;82(1):64-73. doi: 10.1111/bcp.12929. Epub 2016 May 2. PMID 26972584
- [Background] Yi S, Kim SE, Park MK, Yoon SH, Cho JY, Lim KS, Shin SG, Jang IJ, Yu KS. Comparative pharmacokinetics of HD203, a biosimilar of etanercept, with marketed etanercept (Enbrel(R)): a double-blind, single-dose, crossover study in healthy volunteers. BioDrugs. 2012 Jun 1;26(3):177-84. doi: 10.2165/11631860-000000000-00000. PMID 22515513
- [Background] Davatchi F, Jamshidi AR, Banihashemi AT, Gholami J, Forouzanfar MH, Akhlaghi M, Barghamdi M, Noorolahzadeh E, Khabazi AR, Salesi M, Salari AH, Karimifar M, Essalat-Manesh K, Hajialiloo M, Soroosh M, Farzad F, Moussavi HR, Samadi F, Ghaznavi K, Asgharifard H, Zangiabadi AH, Shahram F, Nadji A, Akbarian M, Gharibdoost F. WHO-ILAR COPCORD Study (Stage 1, Urban Study) in Iran. J Rheumatol. 2008 Jul;35(7):1384. Epub 2008 May 1. PMID 18464299
- [Background] Kawai S, Sekino H, Yamashita N, Tsuchiwata S, Liu H, Korth-Bradley JM. The comparability of etanercept pharmacokinetics in healthy Japanese and American subjects. J Clin Pharmacol. 2006 Apr;46(4):418-23. doi: 10.1177/0091270006286435. PMID 16554449